CLINICAL TRIAL: NCT07242807
Title: Evaluation of Clinical and Functional Outcomes After Minimally Invasive Prostate Interventions: A Multicenter Prospective REDCap Registry (MIST Study)
Brief Title: Minimally Invasive Prostate Interventions Registry (MIST Study)
Acronym: MIST
Status: Not yet recruiting | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other); Medical University of Graz (Other); Hannover Medical School (Other)
Responsible Party: Principal Investigator, Selim Soyturk, Urologist / Coordinating Investigator, Necmettin Erbakan University
Other Study IDs: ReScore25-1
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-11

CONDITIONS: Benign Prostatic Hyperplasia (BPH); Minimal Invasive Surgery; LUTS
Keywords: MIST; Minimally Invasive Surgical Therapy; Rezum; UroLift; Aquablation; Prostatic Artery Embolization; iTind; TPLA; Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 72 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MIST_Cohort: Men aged ≥40 years undergoing minimally invasive prostate interventions (Rezum, Urolift, Aquablation, PAE, iTind, TPLA, TUNA, TUMT) as part of routine clinical care. All participants are observed prospectively in a single registry cohort without assignment to treatment.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Participants receive standard-of-care minimally invasive prostate interventions determined by their treating clinicians. The study does not assign or alter any treatment; it only observes outcomes.

SUMMARY:
This study is a multicenter prospective patient registry designed to evaluate clinical, functional, and safety outcomes after minimally invasive prostate interventions (MIST) performed for benign prostatic obstruction (BPO) secondary to benign prostatic hyperplasia (BPH). The interventions included in this registry represent standard-of-care treatment options and may include Rezum water vapor therapy, UroLift prostatic urethral lift, Aquablation, prostatic artery embolization (PAE), iTind, transperineal laser ablation (TPLA), transurethral needle ablation (TUNA), and transurethral microwave therapy (TUMT).

The registry collects standardized data using a secure REDCap platform from participating international centers. Data elements include demographic characteristics, comorbidities, medication use, laboratory parameters, prostate volume assessments, uroflowmetry, post-void residual measurements, patient-reported symptom scores, sexual function assessments, intraoperative details, complications (classified using Clavien-Dindo), and postoperative recovery parameters. Follow-up visits occur at 1, 3, 6, 12, 24, and 36 months, with an optional extended follow-up at 72 months to assess long-term durability and reintervention-free survival.

The primary aim of the study is to evaluate improvements in urinary symptoms (IPSS), quality of life, maximum urinary flow rate (Qmax), and post-void residual volume (PVR) following MIST procedures. Secondary objectives include assessing perioperative safety, catheterization duration, predictors of treatment success or failure, need for reintervention, and long-term preservation of continence and sexual function.

This registry is observational and does not assign or modify any treatment. All procedures are performed based on local clinical practice and physician judgment. Prospective participants provide informed consent. Data collected will be used to generate real-world evidence to guide patient selection, optimize procedural outcomes, and compare clinical performance across different minimally invasive prostate interventions.

DETAILED DESCRIPTION:
Benign prostatic obstruction (BPO) secondary to benign prostatic hyperplasia (BPH) is a prevalent cause of lower urinary tract symptoms (LUTS) in aging men. Minimally invasive surgical therapies (MIST) have become increasingly utilized due to their favorable safety profiles, reduced hospitalization times, preservation of sexual function, and quicker return to normal activities. Despite their growing use, comparative real-world data across MIST modalities remain limited, especially regarding long-term functional outcomes and retreatment rates.

The MIST Registry is an investigator-initiated, non-commercial, multicenter, observational cohort study coordinated by the Department of Urology at Necmettin Erbakan University. The aim is to systematically collect high-quality clinical data from centers using a standardized REDCap electronic data capture system. The registry includes patients treated with any guideline-supported minimally invasive prostate intervention, including Rezum, UroLift, Aquablation, prostatic artery embolization (PAE), iTind, TPLA, TUNA, and TUMT. These procedures are performed as part of routine clinical care and not assigned by the study.

Data collection includes demographics, comorbidities, prior BPO treatments, LUTS medication history, PSA levels, prostate volume, presence and size of median lobe, uroflowmetry parameters, PVR, patient-reported outcomes (IPSS, QoL, IIEF-5, MSHQ-EjD), and urodynamic findings when available. Intraoperative data include type of MIST technique, procedure duration, device usage, energy delivery parameters, imaging guidance, estimated blood loss, and intraoperative complications. Postoperative outcomes include catheterization duration, early complications within 30 days, rehospitalization, urinary retention, infections, and device-related events. Complications are categorized according to the Clavien-Dindo classification, and bladder injury can be scored using the BICEP system where relevant.

Follow-up assessments occur at 1, 3, 6, 12, 24, and 36 months, with optional long-term evaluations at 72 months. Outcomes assessed include symptom scores, Qmax, PVR, PSA, medication changes, and any surgical or minimally invasive reinterventions. Statistical analyses will include descriptive summaries, longitudinal comparisons, multivariable modeling to identify predictors of success or failure, and Kaplan-Meier estimates of reintervention-free survival.

The registry is designed to generate real-world evidence that reflects routine clinical practice across diverse populations and healthcare systems. Findings are expected to inform patient selection, refine procedural decision-making, improve counseling on expected outcomes, and support comparative effectiveness research among emerging minimally invasive prostate treatments.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged ≥40 years
* Diagnosis of benign prostatic hyperplasia (BPH) with lower urinary tract symptoms (LUTS) or benign prostatic obstruction (BPO)
* Undergoing a minimally invasive prostate intervention (Rezum, UroLift, Aquablation, PAE, iTind, TPLA, TUNA, TUMT) as part of standard clinical care
* Ability and willingness to attend scheduled follow-up visits
* Prospective participants able to provide written informed consent
* Retrospective cases eligible if data are fully de-identified and inclusion is approved by local ethics/IRB authorities

Exclusion Criteria:

* Active urinary tract infection at the time of treatment
* ASA physical status ≥5
* Prior pelvic radiotherapy resulting in severe bladder dysfunction
* Severe cognitive impairment or inability to participate in follow-up
* Missing essential baseline data (for retrospective entries)
* Patients receiving experimental or investigational prostate devices or therapies outside routine clinical care

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men aged 40 years and older undergoing minimally invasive prostate interventions for benign prostatic hyperplasia/lower urinary tract symptoms (BPH/LUTS) or benign prostatic obstruction (BPO) across multiple international centers. All treatments are standard-of-care MIST procedures, and participants are followed longitudinally in a single observational registry cohort.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in International Prostate Symptom Score (IPSS) | Baseline; 1, 3, 6, 12, 24, 36, and optional 72 months post-procedure
  IPSS is a validated 0-35 questionnaire assessing lower urinary tract symptoms. Lower scores indicate symptom improvement. Change from baseline will be evaluated at each follow-up visit using patient-reported scores collected via standardized REDCap forms.
Change in maximum urinary flow rate (Qmax) | Baseline; 1, 3, 6, 12, 24, 36, and optional 72 months post-procedure
  Qmax (mL/s) is measured by uroflowmetry at each clinical visit. Improvement in urinary flow represents treatment effectiveness. Change from baseline will be analyzed longitudinally.
Change in quality of life (QoL) score (IPSS subscore) | Baseline; 1, 3, 6, 12, 24, 36, and optional 72 months post-procedure
  QoL score ranges from 0-6. Lower scores reflect improved quality of life. Change from baseline is measured using the IPSS-QoL item collected through REDCap.

SECONDARY OUTCOMES:
Change in Post-Void Residual (PVR) volume | Baseline; 1, 3, 6, 12, 24, 36, and optional 72 months
  PVR (mL) measured by ultrasound or bladder scanner. Lower values indicate improved bladder emptying.
Change in sexual function (IIEF-5 score) | Baseline; 1, 3, 6, 12, 24, 36, 72 months
  IIEF-5 is a validated 5-item erectile function scale (5-25). Higher scores indicate better sexual function.
Change in ejaculatory function (MSHQ-EjD score) | Baseline; 1, 3, 6, 12, 24, 36, 72 months
  MSHQ-EjD evaluates ejaculatory function and bother. Higher function scores indicate improvement.
Catheterization duration | Within first 30 postoperative days
  Duration of urinary catheter use (days) recorded after MIST procedures.
Early postoperative complications (Clavien-Dindo classification) | Within 30 postoperative days
  Complications will be categorized using Clavien-Dindo Grade I-V based on standardized definitions.
BICEP bladder injury score | During the procedure
  Bladder injury is graded using the validated BICEP classification (0-4b). Applicable only when morcellation or bladder instrumentation is performed.
Reintervention rate | Up to 72 months
  Need for additional surgery or MIST (TURP, AEEP/HoLEP, repeat MIST, PAE, Aquablation, urethrotomy, implant revisions, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Selçuk Güven, MD, PhD, Principal Investigator — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University Medical Faculty Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be available upon reasonable request for research purposes. Data will be shared following local ethics committee approval and execution of a data-use agreement. No direct patient identifiers will be shared. Data will include demographic variables, baseline assessments, operative details, postoperative outcomes, and follow-up measures collected in the registry.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data (IPD) and supporting documents will be available beginning 12 months after publication of the primary results manuscript and will remain available for a minimum of 5 years thereafter.
Access Criteria: Only qualified researchers with a methodologically sound proposal will be granted access. Requests must be reviewed and approved by the principal investigator and require completion of a data-use agreement. Access will be provided in de-identified format only and delivered via secure, password-protected electronic transfer. No direct identifiers or protected health information will be shared.

REFERENCES:
- [Background] Rukstalis D, Grier D, Stroup SP, Tutrone R, deSouza E, Freedman S, David R, Kamientsky J, Eure G. Prostatic Urethral Lift (PUL) for obstructive median lobes: 12 month results of the MedLift Study. Prostate Cancer Prostatic Dis. 2019 Sep;22(3):411-419. doi: 10.1038/s41391-018-0118-x. Epub 2018 Dec 12. PMID 30542055
- [Background] Cornu JN, Zantek P, Burtt G, Martin C, Martin A, Springate C, Chughtai B. Minimally Invasive Treatments for Benign Prostatic Obstruction: A Systematic Review and Network Meta-analysis. Eur Urol. 2023 Jun;83(6):534-547. doi: 10.1016/j.eururo.2023.02.028. Epub 2023 Mar 22. PMID 36964042
- [Background] Huang SW, Tsai CY, Tseng CS, Shih MC, Yeh YC, Chien KL, Pu YS, Tu YK. Comparative efficacy and safety of new surgical treatments for benign prostatic hyperplasia: systematic review and network meta-analysis. BMJ. 2019 Nov 14;367:l5919. doi: 10.1136/bmj.l5919. PMID 31727627